CLINICAL TRIAL: NCT03741894
Title: Examination of the Prevention and Treatment Modalities of Alveolitis in Relation With Impacted Teeth Surgery
Acronym: AITS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Pecs (Other)
Responsible Party: Principal Investigator, Balazs Soos, DMD, Assistant Professor, University of Pecs
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 7065-PTE 2018.
Record Dates: First submitted 2018-10-30; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Alveolitis of Jaw; Alveoli, Teeth; Inflammation; Dry Socket; Impacted Third Molar Tooth
Keywords: alveolitis; iodoform; chlorhexidine; minor complications
MeSH Terms: conditions — Dry Socket; Inflammation | interventions — iodoform; Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Primary wound closure (Placebo Comparator): Routine primary wound closure with single interrupted sutures (Surgilon 3-0 non-absorbable) only.
  Interventions: Other: Wound closure using sutures
- Iodoform and wound closure (Experimental): Patients get iodoform (1000 grams containing 350 grams of iodoform, 300 grams of glycerin and 350 grams of alcohol 96%) soaked gauze (steril selvedge gauze bandage 2 cm x 5 m in appropriate length) drainage during suture (Surgilon 3-0 non-absorbable) placements for a week.
  Interventions: Drug: Iodoform; Other: Wound closure using sutures
- Chlorhexidine and wound closure (Experimental): Extraction sockets are filled with 1% chlorhexidine gel (Curasept ADS310, Sager Pharma, Sager Dental Kft.,Budapest, Hungary) before suture (Surgilon 3-0 non-absorbable) placements.
  Interventions: Other: Wound closure using sutures; Drug: Chlorhexidine

INTERVENTIONS:
Drug: Iodoform — Patients get iodoform (1000 grams containing 350 grams of iodoform, 300 grams of glycerin and 350 grams of alcohol 96%) soaked gauze (steril selvedge gauze bandage 2 cm x 5 m in appropriate length) drainage during suture placements for a week.
  Arms: Iodoform and wound closure
Other: Wound closure using sutures — Routine primary wound closure with single interrupted sutures (Surgilon 3-0 non-absorbable) only.
Drug: Chlorhexidine — Extraction sockets are filled with 1% chlorhexidine gel (Curasept ADS310, Sager Pharma, Sager Dental Kft.,Budapest, Hungary) before suture (Surgilon 3-0 non-absorbable) placements.
  Arms: Chlorhexidine and wound closure

SUMMARY:
In the everyday clinical practice the incidence of minor complications is approximately 15-20% of the total number of third molar removals. Alveolitis (dry socket syndrome) may arise in 30-40% of the surgical tooth removals. Several preventive approaches are known, such as the use of iodoform gauze, zink-oxide eugenol paste, platelet rich fibrin (PRF), different medicine containing pastes, like antibiotics containing, non-steroid pain killer containing, steroid containing, or the application of chlorhexidine gel and solutions. In the case of a manifest alveolitis these methods can be used as well. The aims of this research are: i) to identify the important pathogens which play role in the development of alveolitis (microbiological methods), ii) to analyze the in vitro effectivity of the different antiseptic materials in case of infections (inhibitory zones) iii) to compare the effectivity of different alveolitis preventive methods in a prospective clinical study, iv) to compare the different treatment options in alveolitis in a prospective clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Pell-Gregory II/B impaction
* mesioangular impactions
* tooth sectioning is not necessary for removal
* without local infection of third molar

Exclusion Criteria:

* no general diseases or following treatments (DM, steroids, bleeding risk, chemotherapy, radiotherapy, bisphosphonates, immunosuppressive conditions)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in minor postoperative complications (trismus) | day of surgery, 3rd, 7th postoperative days
  Measuring postoperative trismus (maximal mouth opening - inter-incisal distance in millimeters).
Change in minor postoperative complications (oedema) | day of surgery, 3rd, 7th postoperative days
  measuring postoperative oedema (flexible ruler- lateral canthus-mandibular angle distance in millimeters and tragus-labial commissure distance in millimeters).
Change in minor postoperative complications (pain) | 1st, 2nd, 3rd, 4th, 5th, 6th and 7th postoperative days
  Measuring level of pain in Visual Analog Scale (minimum score is 0 which represents no pain, maximum score is 10 which shows the worst pain) postoperatively
Change in necessity of postoperatively taken analgesics | 1st, 2nd, 3rd, 4th, 5th, 6th and 7th postoperative days
  Registering dose of active agent of taken analgesics in milligrams .
Change in necessity of postoperatively taken analgesics | 1st, 2nd, 3rd, 4th, 5th, 6th and 7th postoperative days
  Registering number of daily repeats of taken analgesics.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Oral and Maxillofacial Surgery, University of Pécs, Pécs, Hungary

IPD SHARING:
Plan to Share IPD: Undecided